CLINICAL TRIAL: NCT00834041
Title: An 8-day Open-label, Multiple-dose, Multicenter Study to Evaluate the Safety/Tolerability and Pharmacokinetics of Aliskiren in Hypertensive Pediatric and Adolescent Patients 6-17 Years of Age
Brief Title: A Study to Evaluate the Safety/Tolerability and Pharmacokinetics of Aliskiren in Hypertensive Pediatric and Adolescent Patients 6-17 Years of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A2256
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: aliskiren; pediatric; hypertension; pharmacokinetics (PK); pharmacodynamics (PD); plasma renin activity; mini-tablet formulation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren 2 mg/kg (Experimental): Oral mini-tablets (3.125 mg) of aliskiren dosed at 2 mg/kg body weight once each morning
  Interventions: Drug: Aliskiren 3.125 mini-tablets
- Aliskiren 6 mg/kg (Experimental): Oral mini-tablets (3.125 mg) of aliskiren dosed at 6 mg/kg body weight once each morning
  Interventions: Drug: Aliskiren 3.125 mini-tablets

INTERVENTIONS:
Drug: Aliskiren 3.125 mini-tablets — Oral mini-tablets (3.125 mg) of aliskiren once each morning

SUMMARY:
This first open-label study in a pediatric population was designed to evaluate aliskiren safety and pharmacokinetics after single and multiple dosing in 6-17 year old children with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 6-17 years of age
* Documented history of hypertension as defined in National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents (2004)
* Must be ≥ 21.0 kg and ≤ 100.0 kg at randomization
* Able to safely wash out previous antihypertensive therapy for 1-2 weeks

Exclusion Criteria:

* Body weight of < 21 kg (45 lbs) or > 100 kg (220 lbs)
* Inability to discontinue prior antihypertensive medication as required during the washout period
* Any clinically significant abnormalities or clinically noteworthy abnormal laboratory values
* Renal artery stenosis
* Current diagnosis of heart failure (NYHA Class II-IV)
* msSBP ≥ 25% above the 95th percentile for age, gender, and height at Visit 2
* Second or third degree heart block with or without a pacemaker
* Atrial fibrillation or atrial flutter at Visit 1, or potentially life threatening or any symptomatic arrhythmia during the 12 months prior to Visit 1
* Evidence of current symptomatic valvular disease

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (5):
- Investigative Site, Louisville, Kentucky, United States
- Investigative Site, Brussels, Belgium
- Investigative Site, Brasília, Brazil
- Investigative Site, Budapest, Hungary
- Investigative Site, Warsaw, Poland

REFERENCES:
- [Derived] Sullivan JE, Keefe D, Zhou Y, Satlin L, Fang H, Yan JH. Pharmacokinetics, safety profile, and efficacy of aliskiren in pediatric patients with hypertension. Clin Pediatr (Phila). 2013 Jul;52(7):599-607. doi: 10.1177/0009922813483875. Epub 2013 Apr 22. PMID 23610239

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren 2 mg/kg: Patients received aliskiren 2 mg/kg of their body weight orally once daily at approximately 8 AM.
- Aliskiren 6 mg/kg: Patients received aliskiren 6 mg/kg of their body weight orally once daily at approximately 8 AM.
Period: Overall Study
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg
Started | 19 | 20
Completed | 18 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg | Total
Number analyzed (Participants) | 19 | 20 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 12.2 (3.12) | 11.8 (3.78) | 12.0 (3.44)
Age, Customized [Number; unit: participants]
  6-11 years old | 10 | 10 | 20
  12-17 years old | 9 | 10 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) at Day 1 and Day 8 in 6-11 and 12-17 Year Old Patients
Description: Blood samples (1 mL) for pharmacokinetic (PK) evaluation were drawn pre-dose and at 0.5, 1, 1.5, 2, 3, 4, 6, 10, and 24 hours following administration of aliskiren on Day 1 and Day 8. The pre-dose PK evaluations were collected in a fasted state (7-12 hours without food or beverage except water). PK parameters were calculated from plasma concentration-time data and actual recorded sampling times for each patient, using non-compartmental methods with the software program WinNonlin Pro v5.2.
Time Frame: Day 1 and Day 8
Population: Pharmacokinetic population: All patients who had evaluable aliskiren concentration data.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg
Number analyzed (Participants) | 19 | 20
ng/ml
  Day 1: 6-11 years old, n=10, 10 | 76.8 (78.21) | 393.3 (377.37)
  Day 8: 6-11 years old, n=9, 10 | 82.2 (97.85) | 397.1 (187.06)
  Day 1: 12-17 years old, n=9, 10 | 136.5 (132.57) | 424.3 (188.79)
  Day 8: 12-17 years old, n=9, 10 | 278.7 (357.54) | 485.7 (300.58)

2. Secondary Outcome: Change in Plasma Renin Activity From Baseline on Day 1, Day 8, and Day 9
Description: Blood samples (2 mL) for pharmacodynamics evaluation of plasma renin activity were drawn pre-dose and at 2 and 10 hours following the dose of study medication on Day 1 and at pre-dose and at 2, 10, and 24 hours post-dose on Day 8-9.
Time Frame: Baseline to 2 and 10 hours post-dose on Day 1; pre-dose, 2, 10, and 24 hours post-dose on Day 8-9
Population: Full Analysis Set (FAS): All randomized patients, excluding mis-randomized patients. Data was not available for all patients at all time points. For each time point, n = the number of subjects for whom data was available for each treatment group.
Measure: Mean (Standard Deviation); unit: ng/mL/h
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg
Number analyzed (Participants) | 19 | 20
ng/mL/h
  Day 1: 2 h post-dose, n=15, 15 | -1.8 (1.62) | -4.0 (6.68)
  Day 1: 10 h post-dose, n=14, 13 | -1.8 (1.73) | -3.8 (6.79)
  Day 8: pre-dose, n=14, 15 | -1.3 (1.77) | -3.5 (5.91)
  Day 8: 2 h post-dose, n=11, 14 | -1.4 (1.60) | -3.6 (6.79)
  Day 8: 10 h post dose, n=13, 15 | -1.7 (1.81) | -3.8 (6.41)
  Day 8-9: 24 h post dose, n=13, 15 | -1.5 (1.82) | -3.6 (6.46)

3. Secondary Outcome: Change in Mean Sitting Systolic and Diastolic Blood Pressure (msSBP and msDBP) From Baseline to the End of Treatment (Day 9) in 6-11 and 12-17 Year Old Patients
Description: Blood pressure (BP) measurements were made with a mercury sphygmomanometer or an automated blood pressure measuring device. Sitting BP was measured 3 times at 2-3 minute intervals after the patient had been sitting for 5 minutes. Means of the 3 measurements were calculated. A negative change in BP indicates lowered BP.
Time Frame: Baseline to end of treatment (Day 9)
Population: Full Analysis Set (FAS): All randomized patients, excluding mis-randomized patients.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg
Number analyzed (Participants) | 19 | 20
mmHg
  msSBP: 6-11 years old, n=10, 10 | -4.5 (14.63) | -7.7 (11.76)
  msSBP: 12-17 years old,n=9, 10 | -7.6 (9.07) | -7.7 (9.38)
  msDBP: 6-11 years old, n=10, 10 | -1.7 (4.69) | 0.0 (8.87)
  msDBP: 12-17 years old, n=9, 10 | -5.3 (8.78) | -5.8 (8.00)

4. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC0-τ) in One Dosing Interval (24 h) at Day 1 and Day 8 in 6-11 and 12-17 Year Old Patients
Description: as for outcome 1
Time Frame: Day 1 and Day 8
Population: Pharmacokinetic population: All patients who had evaluable aliskiren concentration data.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg
Number analyzed (Participants) | 19 | 20
h*ng/mL
  Day 1: 6-11 years old, n=10, 10 | 278.3 (237.29) | 1231.0 (728.46)
  Day 8: 6-11 years old, n=9, 10 | 403.6 (326.76) | 1959.9 (821.43)
  Day 1: 12-17 years old, n=9, 10 | 390.9 (264.50) | 1808.7 (806.78)
  Day 8: 12-17 years old, n=9, 10 | 847.2 (803.44) | 2087.0 (999.10)

5. Primary Outcome: Apparent Plasma Clearance (CL/F) at Day 8 in 6-11 and 12-17 Year Old Patients
Description: as for outcome 1
Time Frame: Day 8
Population: Pharmacokinetic population: All patients who had evaluable aliskiren concentration data.
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg
Number analyzed (Participants) | 19 | 20
mL/h/kg
  Day 8: 6-11 years old, n=9, 10 | 9694.0 (8704.71) | 3905.4 (2628.52)
  Day 8: 12-17 years old, n=9, 10 | 5388.1 (5580.55) | 3539.0 (1587.49)

ADVERSE EVENTS:
Time Frame: 12 days
Arm/Group | Aliskiren 2 mg/kg | Aliskiren 6 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/20
Other Adverse Events (participants affected / at risk) | 10/19 | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 2 mg/kg (N=19) | Aliskiren 6 mg/kg (N=20)
Swine influenza (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren 2 mg/kg (N=19) | Aliskiren 6 mg/kg (N=20)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.